CLINICAL TRIAL: NCT02678819
Title: Use of a Wearable Digital Cognitive Aid in Simulated Anesthesia and Intensive Care Crises.
Acronym: SIMMAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEJKA Jean-Christophe (Other)
Responsible Party: Sponsor-Investigator, CEJKA Jean-Christophe, MD PhD, Claude Bernard University
Organization: Claude Bernard University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMMAX UCBL
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Cognitive Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital Aid (Experimental): The digital cognitive aid is designed as a smartphone app. Intervention : cognitive aid during anesthesia and intensive care crises management.
  Interventions: Device: Digital cognitive aid
- No digital aid (No Intervention): Anesthesia and intensive care crises managed without any cognitive aid.

INTERVENTIONS:
Device: Digital cognitive aid — Digital cognitive aid during anesthesia and intensive care crises.
  Arms: Digital Aid

SUMMARY:
The purpose of this study is to determine whether a wearable digital cognitive aid has an effect in the management of simulated crises in anesthesia or intensive care.

DETAILED DESCRIPTION:
" Errare humanum est ", to err is human. This Latin saying attributed to Seneca shows that since the dawn of time, human beings are aware that managing complex situations will always be an inexhaustible source of mistakes. This is particularly true in anesthesia and intensive care in which situations are often complex and stressful, thus leading to mistakes or inadequate management. Improvement might arise from the use of cognitive aids.

The investigators designed a smartphone application including 5 scenarios of anesthesia and intensive care crises (malignant hyperthermia, anaphylactic shock, acute toxicity of local anesthetics, severe and symptomatic hyperkaliemia, ventricular fibrillation), easy to use with a manual validation of every simple step. Investigators seek to compare the technical and non technical management of these crises with and without this wearable cognitive aid.

ELIGIBILITY:
Inclusion Criteria:

* Resident Physicians training in Anesthesia/Intensive care (same specialization in France), year 2 to 5 (out of 5)

Exclusion Criteria:

* All other residents, including Resident Physicians training in Anesthesia/Intensive care, year 1 (out of 5)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Technical Performance as compared to a Reference Task List | Time 0-30 min
  Number of tasks successfully performed, rated on remote video review

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe CEJKA, MD PhD mEng, Principal Investigator — Centre Lyonnais d'Enseignement par la Simulation en Santé, LYON
Locations (1):
- Centre Lyonnais d'Enseignement par la Simulation en Santé, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lelaidier R, Balanca B, Boet S, Faure A, Lilot M, Lecomte F, Lehot JJ, Rimmele T, Cejka JC. Use of a hand-held digital cognitive aid in simulated crises: the MAX randomized controlled trial. Br J Anaesth. 2017 Nov 1;119(5):1015-1021. doi: 10.1093/bja/aex256. PMID 29028930